CLINICAL TRIAL: NCT00205608
Title: Microglia Activation in Schizophrenia: a Pilot Study
Brief Title: Microglia Activation in Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: UMC Utrecht (Other)
Responsible Party: B.N.M. van Berckel, VU Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2002/194
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2008-07

CONDITIONS: Schizophrenia
Keywords: schizophrenia; microglia; PET
MeSH Terms: conditions — Schizophrenia | interventions — Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Positron Emission Tomography — camera is new
  Other Names: Siemens HR+

SUMMARY:
Patients with schizophrenia have volume loss in gray matter. This study is designed to evaluate whether their is microglia activation in schizophrenia using [11C](R)-PK11195 PET.

DETAILED DESCRIPTION:
Schizophrenia is a complex and chronic disease that affects different aspects of cognition and behaviour, including attention, perception, thought processes, emotion and volition. Schizophrenia is a brain disease particularly involving decrement in gray matter as has been supported by findings from many imaging studies. The pathophysiology of these gray matter changes has not been clarified. Microglia activation is the consequence of virtually all conditions associated with neuronal injury. When activated following neuronal damage, microglia show a marked increase in the expression of peripheral type benzodiazepine binding sites which are particularly abundant on cells of the mononuclear macrophage.

(R)-PK11195 [1-(2-chlorophenyl)-N-methyl-N-1(1-methylpropyl]-3 isoquinolinecarboxamide) is a highly selective ligand for the peripheral benzodiazepine binding site. (R)-PK11195, labelled with the positron emitter carbon-11, can be used to monitor the peripheral type benzodiazepine receptors using Positron Emission Tomography (PET). At the Vrije Universiteit Medical Centre (R)-[11C]PK11195 is used for studying microglia activation in-vivo in patients with traumatic brain damage, minimal cognitive impairment and Alzheimer disease.

The objective of this study is to determine whether and to what extent microglia activation occurs in schizophrenia. Ten patients with schizophrenia will be recruited and 10 controls, matched for age and gender. This is an open study. The study consists of one PET scan, which will be performed at the Clinical PET Centre of the Vrije Universiteit Medical Centre. All subjects will also get a MRI scan, which will be performed at the department of Radiology, University Medical Centre Utrecht.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia according to DSM-IV criteria confirmed by a diagnostic interview (CASH, only for patients) within the first 5 years after initial diagnosis
* Male and Females
* Good physical or mental (controls) Health which will be evaluated with medical history, a physical examination and screening laboratory tests (see appendix 1).
* Age between 18 and 40 years (10 patients and 10 controls)
* Mini Mental State score >27 .
* Written informed consent of the subject.
* Hb must be >8 mmol \ litre at the time of the screening.

Exclusion Criteria:

* Previous neurotrauma with loss of consciousness
* Any clinical significant abnormality of any clinical laboratory test, including drug screening.
* Any subject who has received any investigational medication within 30 days prior to the start of this study, or who is scheduled to receive an investigational drug.

any other major current psychiatric diagnosis on axis-1 of DSM-IV (patients)

* History of psychiatric or neurological illness (controls)
* History of psychiatric or neurological illness in first-degree relatives (controls)
* History of alcohol and/or drug abuse (DSM-IV criteria)
* Blood donation within 3 months before the scan day
* Claustrophobia
* Metal objects in or around the body (braces, pacemaker, metal fragments); Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-01; Primary Completion 2007-03 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
[11C]-(R)-Pk11195 binding | within 5 years of start symptoms
  microglia activation in schizophrenia

CONTACTS AND LOCATIONS:
Overall Officials: Bart van Berckel, MD; PhD, Principal Investigator — UMC Utrecht
Locations (1):
- VU University Medical Center, Amsterdam, Amsterdam, Netherlands